CLINICAL TRIAL: NCT05742698
Title: Double Blind Crossover Clinical Trial of Nabilone for Agitation in Frontotemporal Dementia
Brief Title: Nabilone for Agitation in Frontotemporal Dementia
Acronym: Nabilone-FTD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Simon Ducharme, MD (Other)
Collaborators: Alzheimer's Drug Discovery Foundation (Other)
Responsible Party: Sponsor-Investigator, Simon Ducharme, MD, Associate Professor, McGill University, Douglas Mental Health University Institute
Organization: Douglas Mental Health University Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Nabilone-FTD
Record Dates: First submitted 2022-11-23; First posted 2023-02-24 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Frontotemporal Dementia; Frontotemporal Dementia, Behavioral Variant; Primary Progressive Aphasia; bvFTD; PPA; FTD
Keywords: Nabilone; Nabilone FTD; Agitation; TEVA Nabilone; Dementia; BvFTD; FTD
MeSH Terms: conditions — Frontotemporal Dementia; Pick Disease of the Brain; Aphasia, Primary Progressive; Psychomotor Agitation; Dementia | interventions — nabilone

STUDY DESIGN:
Intervention Model Description: This is a multi-centre double blind, placebo-controlled randomized cross-over study comparing 6 weeks of nabilone treatment to 6 weeks of placebo with a 3-week washout between periods. The study will involve an established network of up to 8 FTD centres in Canada.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized using variable block sizes concealed from participating sites. Central randomization will be done with the database and project manager software, REDCap.
  After consent and screening, study staff will enter disease severity into the electronic data capture system randomization module so the research pharmacist will be notified via email of study ID and disease severity. Participants will be randomly assigned to receive either Nabilone or placebo for the first treatment phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nabilone (Active Comparator): Weeks 1-2 Nabilone and placebo will be taken orally by the patient as per the schedule provided by the research team. All patients will start with one 0.5mg capsule per day, taken before bed for the first week and then increase administration to the 1mg capsule taken before bed for the second week.
  Weeks 3-4 Two weeks after the start of the trial patients and study partners will attend an in person or remote Interim Assessment. If remission is not achieved and no clinically significant adverse drug reactions are reported then the dose schedule will increase to 2 capsules per day (2mg/day), 1 capsule in the morning and 1 before bed.
  Weeks 5-6 Four weeks after the start of the trial there will be a second in person or remote Interim Assessment identical to the first. If remission of agitation has not been achieved and no adverse drug reactions are reported the dose schedule will increase to 4 tablets per day (4mg/day), with 2 tablets in the morning and 2 before bed.
  Interventions: Drug: Nabilone
- Placebo (Placebo Comparator): Weeks 1 and 2 Participants will receive one capsule per day to be taken orally before bedtime.
  Weeks 3-4 Participants will receive 2 capsules per day, one in the morning and one before bedtime.
  Weeks 5-6 Participants will receive 2 capsules per day, one in the morning and one before bedtime.
  The placebo dosing regimen is designed to be as similar as possible to the nabilone dosing regime, including using identical capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nabilone — Nabilone is a synthetic cannabinoid that has shown benefit for agitation in Alzheimer's disease. Nabilone further has potentially beneficial properties on oxidative stress and inflammation in neurodegenerative diseases, mechanisms that have been linked to the pathophysiology of frontotemporal dementia.
  Other Names: Nabilone Oral Capsule; TEVA Nabilone
  Arms: Nabilone
Drug: Placebo — The placebo is a capsule identical to the nabilone capsules that will be used in this clinical trial.
  Arms: Placebo

SUMMARY:
The primary goal of this study is to test the hypothesis that oral nabilone treatment will reduce agitation compared with placebo in patients with Frontotemporal Dementia (both behavioural variant frontotemporal dementia and primary progressive aphasia). The study population is defined as patients with probable Frontotemporal Dementia that meet the International Psychogeriatric Association criteria for agitation in cognitive disorders.

DETAILED DESCRIPTION:
While the search for disease modifying treatment of frontotemporal dementia (FTD) remains elusive, on a day-to-day basis, clinicians struggle to help manage the severe neuropsychiatric symptoms of FTD. Agitation, irritability and aggression are common features of the behavioral variant of FTD and to a lesser extent in primary progressive aphasia, and these symptoms are strongly linked to care partner burden. Unfortunately, current pharmacological options for neuropsychiatric symptoms have limited efficacy. Agitation, aggressive behaviors and irritability in FTD are usually pharmacologically managed with a trial-and-error approach using a combination of trazodone, selective serotonin reuptake inhibitors, antiepileptic drugs, memantine and frequently, antipsychotics. Unfortunately, current pharmacological treatment options for neuropsychiatric symptoms of FTD have limited efficacy and are often based on small case studies or anecdotal evidence. Trazodone has the most support from randomized control trials, but shows limited effectiveness. Therefore, in clinical practice second-generation ('atypical') antipsychotics are commonly used despite a paucity of scientific evidence in FTD. This practice is problematic as antipsychotic use in dementia bears a significant burden of side-effects, including falls, and increased cerebrovascular accidents and mortality. There is a clear need for new treatments using novel mechanisms for neuropsychiatric symptoms in FTD.

One promising candidate is nabilone, a synthetic cannabinoid that has shown benefit for agitation in Alzheimer's disease. Nabilone further has potentially beneficial properties on oxidative stress and inflammation in neurodegenerative diseases, mechanisms that have been linked to the pathophysiology of FTD. We propose to conduct the first randomized clinical trial of nabilone for agitation, irritability, and aggression in FTD to obtain data on real-life effectiveness and tolerability. There is a need to obtain data on the efficacy of nabilone on a wide variety of neuropsychiatric symptoms beyond agitation in FTD, while also ensuring the safety of the medication (e.g., is there a detrimental effect on apathy and hyperorality, which are common in FTD). We require data on dosing and tolerability in this population, which is younger on average than Alzheimer's disease subjects from previous studies and therefore may tolerate higher doses of nabilone. The objective of this trial is to obtain robust evidence for the effectiveness and tolerability of nabilone in FTD.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years
* Major neurocognitive disorder due to probable behavioural variant FTD (Rascovsky criteria)17 or primary progressive aphasia (Gorno-Tempini criteria)18. All ages and severity levels will be included.
* Meets International Psychogeriatric Association criteria for agitation in cognitive disorders19
* CMAI score of 39 or above
* Stable psychoactive medication for 2 weeks prior to screening (all medications allowed) with no intention to change dose during treatment period
* Available study partner with ≥10 hours per week in-person contact with the patient. This can either be a friend/family member or a staff member at an assisted living facility.
* Capacity to provide written consent in English or French, or consent from official surrogate decision maker in case of incapacity

Rationale for Inclusion Criteria: The inclusion criteria are designed to enroll patients with FTD with the behaviours of interest, with a range of disease severity that will permit assessment of all outcome measures.

Exclusion Criteria:

* Clinically significant psychotic symptoms (Neuropsychiatric Inventory domain score (severity x frequency) ≥4 on the delusions or hallucinations subscale)
* Clinically significant orthostatic hypotension (a decrease in systolic blood pressure of 20 mm Hg or in diastolic blood pressure of 10 mm Hg within three minutes of standing compared to blood pressure in a seated position)
* Symptomatic orthostatic tachycardia (heart rate increase from of at least 30 beats per minute within the first 5 minutes of standing compared to a seated position IF orthostatic hypotension is not a problem)
* Unstable cardiovascular condition in the opinion of the investigator
* Known or suspected history of drug or alcohol dependence or abuse in the past 12 months, including use of any psychomimetic drugs (e.g. ketamine, lysergic acid diethylamide, psilocybin).
* Allergy, or significant adverse reaction to cannabinoids. If the adverse reaction involved psychological symptoms that are indicative of psychosis or severe anxiety the patient will be excluded. Their treating clinician may be consulted for a clinical opinion on the severity of the response to cannabis and whether this justifies exclusion from the trial.
* Major depressive episode within 6 months of screening
* Women who are breast feeding or pregnant
* Severe liver dysfunction, as determined by their treating clinician
* Other psychiatric or neurological condition that could cause significant agitation
* Ongoing use of any cannabinoid-related products. This includes any THC or CBD based products, regardless of administration method (oral, inhalation, topical, etc…)

Rationale for Exclusion Criteria: The exclusion criteria are designed to avoid inclusion of patients who may have medical comorbidities that would increase their risk of serious side effects from repeated nabilone administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Cohen Mansfield Agitation Inventory (CMAI) | The patients CMAI score will be compared between their Baseline Assessment (prior to starting treatment) and the outcome Assessment (after 6 weeks of treatment) to determine whether agitation has changed across the treatment period.
  A scale that is completed by a caregiver with at lest 10 hours of weekly contact with the patient. This scale evaluates a range of symptoms that fall into the category of agitation.

SECONDARY OUTCOMES:
Tumor necrosis factor alpha (TNFα) | Is TNFα associated with CMAI scores at baseline or with change in CMAI scores after 6-weeks of nabilone treatment (i.e. between Baseline and Outcome Assessments)?
  Examine the relationship between TNFα and CMAI scores at baseline and following nabilone treatment.
4-hydroxynonenal (4-HNE) | Is 4-HNE associated with CMAI scores at baseline or with change in CMAI scores after 6-weeks of nabilone treatment (i.e. between Baseline and Outcome Assessments)?
  Examine the relationship between 4-HNE and CMAI scores at baseline and following nabilone treatment.

OTHER OUTCOMES:
Adverse drug reaction (ADR) to varying doses of nabilone | Count the number of adverse drug reactions that occur accross the 6 week nabiolne treatment period to determine how well this medication is tolerated in this patient population.
  Quantify the prevalence of ADR that occur in response to varying doses of nabilone treatment in patients diagnosed with Frontotemporal Dementia.

CONTACTS AND LOCATIONS:
Locations (7):
- Canada (7):
  - University of British Columbia, St Paul's Hospital, Vancouver, British Columbia
  - Brain and Mind Institute, University of Western Ontario, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Baycrest Hospital, University of Toronto, Toronto, Ontario
  - Western Hospital - University of Toronto, Toronto, Ontario
  - CHU de Québec, Université Laval, Laval, Quebec
  - The Douglas Research Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No
Data will be accessed by members of this multisite research team only, and only de-identified, not individual participant data, will be available to the research team.